CLINICAL TRIAL: NCT03071562
Title: A Randomized Pilot Trial Evaluating the Impact and Feasibility of a Yoga-Mindfulness Intervention on Cognition, Quality of Life, Balance, Walking Speed, Medication Adherence, and Depression in Older Adults Infected With HIV
Brief Title: A Randomized Pilot Trial Evaluating the Impact of a Yoga Intervention on Cognition in Older Adults Infected With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adria Quigley (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Adria Quigley, PhD Student, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4190yogaHIVcog; 371452 (Other Grant/Funding Number: 2016-06-28 Catalyst Grant: HIV/AIDS Community Based Research)
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: HIV/AIDS; Cognitive Impairment; Aging; Mobility Limitation; Medication Adherence; Depression; Quality of Life; Balance Problems
Keywords: HIV; Cognitive impairment; Aging; Physical Activity; Exercise; Yoga; Neuroplasticity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cognitive Dysfunction; Mobility Limitation; Medication Adherence; Depression; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Cognition, motor function (balance, walking speed), and affective (mental health, quality of life, medication adherence) evaluations will be administered at baseline and post-intervention (12 weeks) by a trained physiotherapist, blinded to the group assignment. The rationale for blinding the assessing physiotherapist is to reduce bias in scoring during the outcome assessment sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga-mindfulness (Experimental): Groups of 4-5 participants will engage in group-based sessions supervised by yoga-certified physiotherapists, 60 minutes per intervention/session, 3 sessions/week for 12 weeks. The yoga-mindfulness group will participate in a 60-minute Hatha-style yoga class, with meditation, active postures for strengthening and balance, and breathing exercises. Participants will be tracked for total distance and steps per day using accelerometers (Fitbit Flex).
  Interventions: Other: Yoga-mindfulness
- Control (No Intervention): Participants in this group will not participate in an exercise program. They will be tracked for total distance and steps per day using accelerometers (Fitbit Flex).

INTERVENTIONS:
Other: Yoga-mindfulness — Sample class:
  Warm-up
  (15 minutes) Standing poses
  (15 minutes) Balance poses
  (15 minutes) Abdominals & back bends (10 minutes) Cool-down
  (5 minutes) Seated meditation Alternate nostril breathing Bellows breath Shoulder/neck stretches Cat-cow Forward fold Sun salutations Warrior 1 Warrior 2 Triangle Extended side angle Reverse warrior High lunge with twist Tree pose Standing holding knee Modified warrior 3 (chair support) Half moon
  Bird-dog Side plank Bridge Cobra Sphinx Corpse pose Side-lying Seated om
  Every month, a smudging ceremony will take place with an Aboriginal Elder for 5-10 minutes at the start of the class.
  Arms: Yoga-mindfulness

SUMMARY:
Approximately 50% of people living with HIV (and as many as 80% over the age of 50) have difficulties with cognitive functions such as memory and thinking that can have a profound negative impact on activities of daily living and quality of life. Problems with memory and thinking are also associated with forgetting to take anti-retroviral drugs and experiencing challenges to balance, walking and mental health (anxiety and depression). There is increasing evidence that, in the general population, exercise has positive effects on cognition, physical functioning and mental health. Despite the recognition of multiple therapeutic benefits of exercise, little attention has been paid to its possible effects on cognition in people living with HIV. The purpose of the proposed pilot study is to compare the effects of a 12-week, randomly assigned, community-based yoga-mindfulness intervention on cognition, balance, walking, mental health and quality of life in 30 people >35 years of age living with HIV in the Halifax area. Yoga is of particular interest because it encompasses not only the physical but also spiritual, emotional, and mental dimensions of life. As such, it has tremendous potential to help stave off some of the devastating consequences of HIV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Participant self-report of HIV diagnosis
2. Identified cognitive concerns on the C3Q (Communicating Cognitive Challenges in HIV Questionnaire)
3. Residence in the Halifax area
4. Capacity to provide informed consent
5. Aged 35 or older

Exclusion Criteria:

* If participants present with contraindications to exercise, they will be excluded from the study. If participants have participated in a yoga program within the past 6 months, they will be excluded.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
B-CAM (Brief Cognitive Ability Measure) | Will be assessed at baseline and 12 weeks.
  Cognitive function will be measured using the Brief Cognitive Ability (B-CAM), a computerized cognitive test developed using Rasch Measurement Theory and Analysis that takes 30 minutes to administer.
C3Q (Communicating Cognitive Challenges in HIV Questionnaire) | Will be assessed during screening, baseline, and 12 weeks.
  Self-reported cognition will be assessed using the C3Q (Communicating Cognitive Challenges in HIV Questionnaire).

SECONDARY OUTCOMES:
Feasibility (Post-participation questionnaire) | Assessed at 12 weeks.
  Many domains of feasibility will be assessed using a post-intervention questionnaire with questions related to participant comfort, satisfaction, safety, attendance, and time commitment.
Balance | Assessed at baseline and at 12 weeks.
  Balance will be measured using the Community Balance and Mobility test (CB&M).
Walking Speed | Assessed at baseline and at 12 weeks.
  Walking peed will be measured using the 10-meter walking test because it is a simple, well-recognized global health indicator that can predict survival probability.
Depression | Assessed at baseline and at 12 weeks.
  Depression will be assessed using the Hospital Anxiety and Depression Scale, a self-report questionnaire.
Medication Adherence | Assessed at baseline and at 12 weeks.
  Participants will also be asked about Medication adherence (specifically antiretroviral) using the Simplified Medication Adherence Questionnaire (SMAQ).
Health-related Quality of Life | Assessed at baseline and at 12 weeks.
  Quality of life will be assessed using MOS-HIV, consisting of 10 domains (health perceptions, physical/role/ social functioning, pain, mental health, vitality, health distress, cognitive function, QOL).

CONTACTS AND LOCATIONS:
Locations (1):
- HIV clinic, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quigley A, Brouillette MJ, Gahagan J, O'Brien KK, MacKay-Lyons M. Feasibility and Impact of a Yoga Intervention on Cognition, Physical Function, Physical Activity, and Affective Outcomes among People Living with HIV: A Randomized Controlled Pilot Trial. J Int Assoc Provid AIDS Care. 2020 Jan-Dec;19:2325958220935698. doi: 10.1177/2325958220935698. PMID 32583707
- [Derived] Quigley A, O'Brien KK, Brouillette MJ, MacKay-Lyons M. Evaluating the Feasibility and Impact of a Yoga Intervention on Cognition, Physical Function, Physical Activity, and Affective Outcomes in People Living With HIV: Protocol for a Randomized Pilot Trial. JMIR Res Protoc. 2019 May 21;8(5):e13818. doi: 10.2196/13818. PMID 31115343